CLINICAL TRIAL: NCT02230683
Title: An Open-Label Pilot Trial to Evaluate the Safety, Tolerability and Efficacy of IDN-6556 in Cirrhotic Subjects With Portal Hypertension
Brief Title: A Study of IDN-6556 in Cirrhotic Subjects With Portal Hypertension
Acronym: PH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDN-6556-11
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-10

CONDITIONS: Liver Cirrhosis; Hepatic Cirrhosis; Portal Hypertension
Keywords: Liver Cirrhosis; Hepatic Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IDN-6556 - Overall population (Experimental): Overall evaluable population treated with IDN-6556 25 mg twice daily
  Interventions: Drug: IDN-6556
- IDN-6556 - Subgroup with Baseline HVPG < 12 mmHg (Experimental): Subgroup for patients with Baseline HVPG < 12 mmHg that have been treated with IDN-6556 25 mg twice daily
  Interventions: Drug: IDN-6556
- IDN-6556 - Subgroup Baseline HVPG ≥ 12 mmHg (Experimental): Subgroup for patients with Baseline HVPG ≥ 12 mmHg that have been treated with IDN-6556 25 mg twice daily
  Interventions: Drug: IDN-6556

INTERVENTIONS:
Drug: IDN-6556 — 25 mg BID
  Other Names: emricasan; PF-013491390

SUMMARY:
This is an open-label pilot study to evaluate the safety, tolerability, and efficacy of IDN-6556 in treating portal hypertension in subjects with liver cirrhosis.

DETAILED DESCRIPTION:
Studies in patients with liver disease have demonstrated that cCK18 is elevated in the serum of patients and has been associated with disease severity. Studies have also shown that cCK18 is generally elevated to a higher degree in cirrhosis than in other liver diseases. In addition, increasing stages of cirrhosis from Child-Pugh A, Child-Pugh B to Child-Pugh C are associated with progressively higher levels of caspase cleaved cytokeratin 18. This suggests that apoptosis and caspase activity are associated with the severity of disease. IDN-6556 and its ability to inhibit inflammation and apoptosis may have a beneficial impact on both the dynamic and structural components associated with the pathogenesis of portal hypertension in cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of minimum adult legal age (according to local laws for signing the informed consent document), able to provide written informed consent, and able to understand and willing to comply with the requirements of the study
* Clinical, radiological, or biochemical evidence of liver cirrhosis
* Evidence of portal hypertension as evidenced by any of the following:

  1. Splenomegaly, on imaging and/or clinical evaluation, with platelet count of <120,000 at study entry, or
  2. Presence of small sized varices on screening endoscopy and/or collateral circulation on imaging, or
  3. Presence of medium/large varices that have never bled and have been obliterated with endoscopic ligation
* Portal hypertension defined as a hepatic venous pressure gradient (HVPG) >5 mmHg at Screening
* Willingness to utilize two reliable forms of contraception (for both males and females of childbearing potential) from Screening to one month after the last dose of study drug.

Exclusion Criteria:

* Decompensated cirrhosis as defined by the presence of overt ascites (requiring diuretics), overt encephalopathy (requiring specific therapy), or history of variceal hemorrhage.
* Known infection with HIV
* Hepatic failure defined as total bilirubin ≥12 mg/dL
* Other non-liver organ failure, including:

  1. Renal failure defined as creatinine ≥ 2.0 mg/dL
  2. Cerebral failure defined as hepatic encephalopathy grade III or IV
  3. Coagulation failure defined as INR ≥ 2.5 or platelets ≤ 20x109/L
  4. Hemodynamic requirement for inotropic support
* Child-Pugh score of 10-15 (Child-Pugh C classification)
* Use of vasoactive drugs (at or within 3 months of Screening) that may impair hepatic blood flow; examples include but are not limited to:

  1. β-blockers, including carvedilol
  2. Nitrates
  3. Vasopressin (or analogues)
  4. Phosphodiesterase inhibitors (prescribed daily for pulmonary hypertension; p.r.n. use for erectile dysfunction is permitted)
* Change in dose or regimen within 3 months of Screening of:

  1. Fibrates or statins
  2. Angiotensin II receptor antagonist or angiotensin converting enzyme (ACE) inhibitor
* Use of the following drugs within 2 months of Screening:

  1. Systemic corticosteroids
  2. Pentoxifylline
  3. Known or suspected use of illicit drugs or drugs of abuse (allowed if medically prescribed or indicated)
* Concomitant pancreatitis
* Evidence of portal vein thrombosis on Doppler ultrasound of the portal vasculature
* Active inflammatory bowel disease
* Diagnosed or suspected systemic lupus erythematosus (SLE) and/or rheumatoid arthritis (RA)
* Autoimmune hepatitis
* Hepatitis C Virus (HCV) infected subjects receiving or planning on receiving anti-viral therapy during the course of the study
* Hepatitis B Virus (HBV) infected subjects who have been on stable anti-HBV therapy for less than 3 months
* Hepatocellular carcinoma (HCC) at entry into the study
* Active non-liver malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas)
* History or presence of clinically concerning cardiac arrhythmias, or prolongation of screening (pre-treatment) QT or QTc interval of >480 milliseconds (msec)
* Significant systemic or major illness other than liver disease, including coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, serious psychiatric disease, that, in the opinion of the Investigator would preclude the subject from participating in and completing the study
* Any subject that has received any investigational drug or device within 30 days of dosing or who is scheduled to receive another investigational drug or device in the course of the study
* If female, known pregnancy, or has a positive urine or serum pregnancy test, or lactating/breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hagerty, MD, Study Chair — Conatus Pharmaceuticals Inc.
Locations (16):
- United States (16):
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Johns Hopkins Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - New York University Lagone Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - St. Luke's Health Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Bon Secours Mary Immaculate Hospital, Newport News, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - McGuire DVAMC, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- IDN-6556: IDN-6556 25 mg Dosed twice daily
Period: Overall Study
Arm/Group | IDN-6556
Started | 23
Completed | 22
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | IDN-6556
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 6
Gender [Count of Participants; unit: Participants]
  Female | 7
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Venous Pressure Gradient (HVPG)
Description: Mean change of HVPG [mmHg] from Baseline to Day 28/EOT (end of treatment) for IDN-6556
Time Frame: Baseline to Day 28/EOT (end of treatment)
Population: 23 subjects were enrolled, of whom 22 were evaluable for the HVPG endpoint. 1 subject discontinued at day 1.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- IDN-6556 - Overall Population: Overall evaluable population treated with IDN-6556 25 mg twice daily with HVPG measurement at Baseline and Day 28
- IDN-6556 - Subgroup With HVPG < 12 mmHg: Subgroup for patients with HVPG < 12 mmHg that have been treated with IDN-6556 25 mg twice daily
- IDN-6556 - Subgroup HVPG ≥ 12 mmHg: Subgroup for patients with HVPG ≥ 12 mmHg that have been treated with IDN-6556 25 mg twice daily
Arm/Group | IDN-6556 - Overall Population | IDN-6556 - Subgroup With HVPG < 12 mmHg | IDN-6556 - Subgroup HVPG ≥ 12 mmHg
Number analyzed (Participants) | 22 | 10 | 12
mmHg
  Baseline | 15.2 (7.68) | 8.05 (1.88) | 20.62 (5.59)
  Day 28/EOT | 14.1 (6.40) | 10.0 (3.86) | 17.6 (6.10)
  Change From Baseline | -1.14 (4.57) | 1.90 (3.15) | -3.67 (4.05)
Statistical Analysis 1: Comparison: IDN-6556 - Overall Population; Statistical Analysis for the mean change of the Hepatic Venous Pressure Gradient from Baseline to Day 28/EOT for the overall evaluable population treated with IDN-6556 25 mg twice daily; Test type: Superiority or Other; p = 0.257, Paired t-test; within group change = -1.14, 95% CI 2-sided [-3.16 to 0.89], Standard Deviation 4.57 — within group change
Statistical Analysis 2: Comparison: IDN-6556 - Subgroup With HVPG < 12 mmHg; Statistical Analysis for the mean change of the Hepatic Venous Pressure Gradient from Baseline to Day 28/EOT in the HVPG < 12 mmHg subgroup; Test type: Superiority or Other; p = 0.1174, ANCOVA; within group change = 1.90, 95% CI 2-sided [-0.52 to 4.32], Standard Deviation 3.15 — within group change
Statistical Analysis 3: Comparison: IDN-6556 - Subgroup HVPG ≥ 12 mmHg; Statistical Analysis for the mean change of the Hepatic Venous Pressure Gradient from Baseline to Day 28/EOT in the HVPG ≥ 12 mmHg subgroup; Test type: Superiority or Other; p = 0.0025, ANCOVA; within group change = -3.67, 95% CI 2-sided [-5.88 to -1.46], Standard Deviation 4.05 — within group change

2. Primary Outcome: cCK18/M30
Description: Absolute Mean Change of caspase-cleaved cytokeratin serum levels (cCK18/M30); the statistical analysis is based on the mean change in log-transformed cCK18/M30 from Baseline to Day 28/EOT (end of treatment) for IDN-6556
Time Frame: Change from Baseline to Day 28/EOT
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- IDN-6556 - Subgroup With HVPG < 12 mmHg: Subgroup for patients with Baseline HVPG < 12 mmHg that have been treated with IDN-6556 25 mg twice daily
- IDN-6556 - Subgroup HVPG ≥ 12 mmHg: Subgroup for patients with Baseline HVPG ≥ 12 mmHg that have been treated with IDN-6556 25 mg twice daily
Arm/Group | IDN-6556 - Overall Population | IDN-6556 - Subgroup With HVPG < 12 mmHg | IDN-6556 - Subgroup HVPG ≥ 12 mmHg
Number analyzed (Participants) | 23 | 10 | 13
U/L | -47.1 (122.23) | -74.3 (99.02) | -26.2 (137.64)
Statistical Analysis 1: Comparison: IDN-6556 - Overall Population; Statistical Analysis for the mean change in log-transformed caspase-cleaved cytokeratin serum levels from Baseline to Day 28/EOT for the overall evaluable population treated with IDN-6556 25 mg twice daily; Test type: Superiority or Other; p = 0.026, ANCOVA; within group change = -0.22, 95% CI 2-sided [-0.42 to -0.03]
Statistical Analysis 2: Comparison: IDN-6556 - Subgroup With HVPG < 12 mmHg; Statistical Analysis for the mean change in log-transformed caspase-cleaved cytokeratin serum levels from Baseline to Day 28/EOT in the HVPG < 12 mmHg subgroup population treated with IDN-6556 25 mg twice daily; Test type: Superiority or Other; p = 0.001, ANCOVA; within group change = -0.46, 95% CI 2-sided [-0.72 to -0.21]
Statistical Analysis 3: Comparison: IDN-6556 - Subgroup HVPG ≥ 12 mmHg; Statistical Analysis for the median change in log-transformed caspase-cleaved cytokeratin serum levels from Baseline to Day 28/EOT in the HVPG ≥ 12 mmHg subgroup population treated with IDN-6556 25 mg twice daily; Test type: Superiority or Other; p = 0.72, ANCOVA; within group change = -0.04, 95% CI 2-sided [-0.26 to 0.18]

3. Primary Outcome: Change in cCK18/M30
Description: Median change of caspase-cleaved cytokeratin serum levels (cCK18/M30) from Baseline to Day 28/EOT (end of treatment) for IDN-6556
Time Frame: Baseline to Day 28/EOT (end of treatment)
Measure: Median (Full Range); unit: U/L
Arm/Group | IDN-6556 - Overall Population | IDN-6556 - Subgroup With HVPG < 12 mmHg | IDN-6556 - Subgroup HVPG ≥ 12 mmHg
Number analyzed (Participants) | 23 | 10 | 13
U/L
  Baseline | 191.0 [78 to 994] | 189.0 [126 to 442] | 221.0 [78 to 994]
  Day 28/EOT | 143.0 [48 to 548] | 124.5 [48 to 291] | 186.0 [94 to 548]
  Change From Baseline at Day 28 | -21.0 [-446 to 119] | -52.5 [-323 to 45] | 12.0 [-446 to 119]
Statistical Analysis 1: Comparison: IDN-6556 - Overall Population; Statistical Analysis for the median change of caspase-cleaved cytokeratin serum levels from Baseline to Day 28/EOT for the overall evaluable population treated with IDN-6556 25 mg twice daily; Test type: Superiority or Other; p = 0.105, Wilcoxon (Mann-Whitney); Hodges-Lehmann = -21, 95% CI 2-sided [-60 to 13]
Statistical Analysis 2: Comparison: IDN-6556 - Subgroup With HVPG < 12 mmHg; Statistical Analysis for the median change of caspase-cleaved cytokeratin serum levels from Baseline to Day 28/EOT in the HVPG < 12 mmHg subgroup population treated with IDN-6556 25 mg twice daily; Test type: Superiority or Other; p = 0.016, Wilcoxon (Mann-Whitney); Hodges-Lehmann = -52.5, 95% CI 2-sided [-109 to -6]
Statistical Analysis 3: Comparison: IDN-6556 - Subgroup HVPG ≥ 12 mmHg; Statistical Analysis for the median change of caspase-cleaved cytokeratin serum levels from Baseline to Day 28/EOT in the HVPG ≥ 12 mmHg subgroup population treated with IDN-6556 25 mg twice daily; Test type: Superiority or Other; p = 0.839, Wilcoxon (Mann-Whitney); Hodges-Lehmann = 12, 95% CI 2-sided [-60 to 13]

4. Secondary Outcome: Change in Alanine Aminotransferase (ALT)
Description: Median change of ALT from Baseline to Day 28/EOT (end of treatment) for IDN-6556
Time Frame: Baseline to 28 days/EOT
Measure: Median (Full Range); unit: U/L
Groups:
- IDN-6556: Overall evaluable population treated with IDN-6556 25 mg twice daily
Arm/Group | IDN-6556
Number analyzed (Participants) | 23
U/L
  Baseline | 25.0 [10 to 99]
  Day 28/EOT | 23.0 [9 to 124]
  Change from Baseline at Day 28 | -4.0 [-61 to 43]
Statistical Analysis 1: Comparison: IDN-6556; Statistical Analysis for the median change in Alanine Aminotransferase (ALT) from Baseline to Day 28/EOT; Test type: Superiority or Other; p = 0.0084, Wilcoxon (Mann-Whitney); Hodges-Lehmann = -4, 95% CI 2-sided [-7 to 0]

5. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: Median change of AST from Baseline to Day 28/EOT (end of treatment) for IDN-6556
Time Frame: Baseline to 28 days/EOT
Measure: Median (Full Range); unit: U/L
Arm/Group | IDN-6556
Number analyzed (Participants) | 23
U/L
  Baseline | 35.0 [16 to 83]
  Day 28/EOT | 27.0 [13 to 139]
  Change from Baseline at Day 28 | -4.0 [-29 to 68]
Statistical Analysis 1: Comparison: IDN-6556; Statistical Analysis for the median change in Aspartate Aminotransferase (AST) from Baseline to Day 28/EOT; Test type: Superiority or Other; p = 0.0131, Wilcoxon (Mann-Whitney); Hodges-Lehmann = -4, 95% CI 2-sided [-7 to -1]

6. Secondary Outcome: Concentration of Caspase 3/7 RLU
Description: Median change of concentration of Caspase 3/7 Relative Light Units from Baseline to Day 28/EOT (end of treatment) for IDN-6556
Time Frame: Baseline to 28 days/EOT
Measure: Median (Full Range); unit: RLU
Arm/Group | IDN-6556
Number analyzed (Participants) | 23
RLU
  Baseline | 1997 [750 to 37428]
  Day 28/EOT | 1518 [276 to 3665]
  Change from Baseline at Day 28 | -772 [-34734 to 1107]
Statistical Analysis 1: Comparison: IDN-6556; Statistical Analysis for the median change in concentration of Caspase 3/7 Relative Light Units from baseline to Day 28/EOT; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney); Hodges-Lehmann = -772, 95% CI 2-sided [-1188 to -19] — The estimated value is the ratio for the difference from baseline

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for a period of 8 months.
Arm/Group | IDN-6556
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (N=23)
Systematic inflammatory response syndrome (General disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (N=23)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 1 (1)
Abdominal disorders (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Local swelling (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 3 (4)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Soft tissue inflammation (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less